CLINICAL TRIAL: NCT03425058
Title: Prospective Study of Molecular Evaluation of Neoadjuvant Chemotherapy for Locally Advanced Gastric Cancer
Brief Title: Molecular Evaluation of Neoadjuvant Chemotherapy for Locally Advanced Gastric Cancer
Acronym: MENCA-GC
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jiafu Ji, Professor, Peking University Cancer Hospital & Institute
Other Study IDs: 2017YJZ38
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Gastric Cancer
Keywords: Molecular Evaluation; Locally Advanced Gastric Cancer; Neoadjuvant Chemotherapy; ctDNA; CTC; dMMR/MSI
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples; formalin-fixed, paraffin-embedded tumor blocks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastric cancer (GC) is a leading global health problem and is the third most common cause of cancer related death. Neoadjuvant chemoradiotherapy (nCRT) followed by surgery is the mainstay treatment for locally advanced gastric cancer, and variable degrees of tumor regression are observed after nCRT. Treatment strategies, including close surveillance without immediate surgery, have been investigated to spare patients with complete tumor regression from potentially adverse outcomes of radical surgery. However, clinical and radiological assessment of treatment response does not deliver an ideal accuracy of patients identification with complete response. In the present study, we focused on the clinical courses of patients who have developed locally advanced gastric cancer, and investigated the potential clinical utility of the detection of deficient MMR(dMMR), microsatellite instability(MSI) status and the decreasing level of circulating tumor cells (CTCs) and circulating tumor DNA (ctDNA) as promising biomarkers for the diagnosis and prediction of GC during treatment progress. Twenty milliliters of plasma were collected at 3 time points: before nCRT; after 2 cycles of nCRT; and after surgery. Firefly ctDNA NGS assays were used to track ctDNA mutations previously characterized in paired tumor tissue by massively parallel sequencing (MPS). We investigated whether circulating tumor DNA (ctDNA) detection can reflect tumor response to nCRT and detect minimal residual disease(MRD) after surgery. We compared CTC and ctDNA levels to clinical, radiological and pathological assessment modalities for nCRT response. The results will provide lots of information which may contribute to promote the treatment of GC patients. We want to introduce these strategies into clinical practice if possible.

DETAILED DESCRIPTION:
This study is a single-center observational study on a patient cohort of at least 80 patients with histologically-confirmed locally advanced gastric cancer (LAGC). The protocol used in this study is approved by the Ethics Committee of Beijing Cancer Hospital.

The primary endpoint is the 3-year progression-free survival (PFS) rate. The secondary endpoints are the overall survival (OS) and safety.

Currently, the best treatment for early and mid-stage LAGC patients is resection but even with successful treatment, most patients still relapse and the 5-year survival rate is less than 30%.

For patients with cT4a/T4bN+M0, including T4b、Bulky-N2, primary lesions are not always fully excised during treatment and prognosis for these patients is generally poor. Recent studies, however, have suggested that the inclusion of neoadjuvant chemotherapy (NCT) can improve patient outcomes by: 1) downstaging tumors and increasing the likelihood of curative resection, 2) reducing the prevalence of micro metastases.

Historically, Oxaliplatin and s-1 combination therapy has been shown to be well-tolerated in patients with recurrent or metastatic gastric cancer.

To best evaluate the treatment response of NCT, we plan to investigate the effect of new technologies and assays on the successful prediction of patient outcomes.

Circulating tumor DNA (ctDNA), fragmented DNA with an average size of 166 bp, is released by cancer cells into circulation. Circulating tumor cells (CTCs) are rare malignant cells detached from tumors which enter the bloodstream. Both these biomarkers can be used for prognosis and the dynamic monitoring of disease progression.

In the MAGIC trial, patients with tumor that are MSI-H or MMRD, had survival rates superior to those with MSS/MSI-L or MMRP tumors when treated with surgery alone.

We will combine dMMR/MSI status with the dynamic evaluation of CTCs and ctDNA using liquid biopsy technology to determine whether changes in tumor burden in response to NTC can identify potential treatment responders.

Sequential peripheral blood samples for CTCs and ctDNA analysis will be taken before and after NCT, as well as one week after surgery.

Tumor assessments will be performed after 2 cycles NCT based on RECIST v1.1 criteria using CT/MRI scan.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory males or females, age ≥ 18 years
2. Karnofsky Performance Score (KPS) ≥70% or ECOG performance status: 0 or 1
3. Pathologically confirmed gastric adenocarcinoma (regardless of degree of histologic differentiation) or adenocarcinoma with signet-ring cell carcinoma , mucinous adenocarcinoma
4. Clinical Preoperative Stage cT4a/T4bN+M0 disease, including T4b、Bulky-N2, confirmed by CT/EUS
5. Adequate organ function as defined below: Hemoglobin ≥ 9 g/dl, Hematologic Absolute Neutrophil Count （ANC） ≥ 1.5*109/L, Platelets ≥ 100*109/L, Aspartate Aminotransferase（AST） and Alanine Aminotransferase(ALT)≤ 2.5×ULN, Alkaline pPosphatase( ALP) ≤ 2.5×ULN, Total Bilirubin （TBIL）≤ 1.5×ULN, Renal Serum Creatinine < 1.5 ULN, Serum Albumin ≥ 30g/l.
6. No serious concomitant disease that make survival period < 5 years
7. No pleural effusion, no ascites exceeding the pelvis and no metastasis to the peritoneum, liver or other distant organs are confirmed by abdominal pelvic CT.
8. Planning to undergo gastric cancer D2 surgery after neoadjuvant chemotherapy
9. No prior antitumor treatment is allowed, including chemotherapy, radiotherapy, immune therapy or target therapy
10. No mechanical obstruction.
11. Negative serum or urine pregnant test within 7 days prior to randomization for child-bearing age women
12. Sexually active males or females willing to practice contraception during the study until 30 days after end of study.
13. Subjects has to voluntarily join the study and sign the Informed Consent Form for the study

Exclusion Criteria:

1. Female in pregnancy or lactation, or refuse to receive Contraception measures during chemotherapy
2. With distant metastasis or peritoneal dissemination diagnosed by CT/EUS
3. Underwent prior antitumor treatment, including chemotherapy, radiotherapy, immune therapy or target therapy
4. Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety (including current active hepatic, biliary, renal, respiratory disease, uncontrolled diabetes hypertension et al)
5. Clinically serious cardiac disease or pulmonary dysfunction.
6. Patients require emergency surgery with complications (bleeding, perforation and obstruction) caused by gastric cancer
7. Other complications that cause no radical resection
8. Serious concomitant disease that make survival period < 5 years
9. No detection of CTCs or ctDNA in peripheral blood samples before NCT be enrolled in other clinical trials
10. Allergic reaction to S-1 or oxaliplatin
11. Abnormal GI tract function
12. Refuse to provide blood/tissue sample
13. Sexually active males or females refuse to practice contraception during the study until 30 days after end of study.
14. Person with no capacity (legally) or inappropriate to continue study treatment for ethics/medical reasons.
15. Other situation to be judged not adaptive to the study by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: locally advanced gastric cancer patients without distant metastasis or peritoneal dissemination defined as cTNM stage of T4a/T4bN+M0
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
The relationship between dMMR/MSI status and response to neoadjuvant chemotherapy | November 22, 2017 to December 31, 2018
  The relationship between dMMR/MSI status and response to neoadjuvant chemotherapy
The concordance and accuracy of response evaluation results determined by ctDNA, CTCs compared with imaging and serum tumor biomarkers(CEA, CA19-9,CA72-4 et al) | November 22, 2017 to December 31, 2018
  The concordance and accuracy of response evaluation results determined by ctDNA, CTCs compared with imaging and serum tumor biomarkers(CEA, CA19-9,CA72-4 et al)

SECONDARY OUTCOMES:
Prognostic values of the CTCs,ctDNA and dMMR/MSI testing | November 22, 2017 to December 31, 2018
  Prognostic values of the CTCs,ctDNA and dMMR/MSI testing
The concordance of mutations in tumor tissue and ctDNA | November 22, 2017 to December 31, 2018
  The concordance of mutations in tumor tissue and ctDNA

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, MD, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China